CLINICAL TRIAL: NCT06591858
Title: Evaluation of Renal Function in Patients With Subclinical and Overt Hyperthyroidism
Brief Title: Evaluation of Renal Function in Patients With Hyperthyroidism
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Khaled Abdelghany, Resident Doctor, Assiut University
Other Study IDs: Hyperthyroidism and kidney
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hyperthyroidism
MeSH Terms: conditions — Hyperthyroidism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the effect of subclinical and overt Hyperthyroidism in renal function

DETAILED DESCRIPTION:
* Thyroid disorders are very common with a high prevalence among the general population. Thyroid diseases are associated with many detrimental effects that have a serious impact on various body systems.(1)

  * Hyperthyroidism can be overt or subclinical. Overt hyperthyroidism is defined as low serum thyroid stimulating hormone (TSH) and elevated serum thyroxin (T4), tri-iodothyronine (T3), or both. Whereas subclinical hyperthyroidism (SCH) is defined as low serum TSH level with normal serum levels of T3 and T4.(2)
  * The relationship between thyroid hormones and kidney function is well-known for many years. Thyroid diseases adversely affect renal physiology; meanwhile, kidney diseases could result in thyroid dysfunction.
* Thyroid hormones contribute to the maintenance of water and electrolyte balance, and participate in the renal transport system. Hyperthyroidism results in an increased glomerular filtration rate (GFR) by about 18-25%. due to increased renal blood flow and activation of renin angiotensin-aldosterone system (RAAS). Also, these changes have been reported in patients with hyperthyroidism.(3-5)
* Several mechanisms were found playing roles on increasing both the size and functional capacity of kidney:

  1. Thyroid hormone directly influences the expression and activity of most of renal transporters by direct binding of thyroid hormone to the promoter region of a transporter gene (6)
  2. In hyperthyroid state beta-adrenergic receptors in kidney cortex, and synthesis and secretion of renin by juxtaglomerular cells are increased, which in turn enhance angiotensin-converting enzyme activity.(7)
  3. Increased RAAS activity results in afferent arteriolar vasodilatation and efferent arteriolar vasoconstriction with a consequent increase in the filtration pressure...(8) D) Hyperthyroidism increases systolic blood pressure by increasing heart rate, decreasing systemic vascular resistance, raising cardiac output, and increases nitric oxide production which all contributes to the hyper dynamic circulation. Hyperthyroidism results in increased renal blood flow.(7)
* Observed that both BUN and creatinine levels increased significantly after euthyroidism was achieved in hyperthyroid patients, these findings point out to true decline in renal function rather than a mere adaptation to hemodynamic changes.

Although the mechanistic link between thyroid and kidney disease remains unclear, hyperthyroidism may have significant effect on renal function

ELIGIBILITY:
Inclusion Criteria:

* Patients aged (18_80 years) diagnosed subclinical and overt Hyperthyroidism with overt Hyperthyroidism

Exclusion Criteria:

1. Patients with D.M
2. Patients with Hypertension
3. Patients with CKD or ESRD
4. IHD
5. Pateints receiving medication known to affect renal function as contrast agent, non-steroidal anti-inflammatory drugs and ACEIs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with overt Hyperthyroidism ( clinically manifested and laboratory by low TSH, high fT3 & fT4) And subclinical hyperthyroidism ( low TSH <0.4.MI/IU without clinical symptoms of hyperthyroidism
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Evaluation of renal function in patients with subclinical and overt Hyperthyroidism. | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed K Abdelghany, Principal Investigator — Assiut University; Hanaa M Riad, Study Director — Assiut University